CLINICAL TRIAL: NCT01669265
Title: Sentinel Lymph Node Total Tumoral Load as a Predictor of Non Sentinel Node Involvement in Early Breast Cancer
Acronym: SOLO-1
Status: Completed | Type: Observational
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Sysmex America, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SOLTI-1113
Record Dates: First submitted 2012-05-24; First posted 2012-08-20 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer; OSNA; sentinel lymph node
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OSNA: Patient cases with cT1-3, N0 early breast cancer, who previously had intraoperative sentinel lymph node (SLN) evaluation by one-step nucleic acid amplification (OSNA) assay with a complete axillary dissection.

SUMMARY:
This is a retrospective, multicentric cohort study of patient cases with cT1-3, N0 early breast cancer, who previously had intraoperative sentinel lymph node (SLN) evaluation by one-step nucleic acid amplification (OSNA) assay with a complete axillary dissection.

The aim of the present study is to assess the intraoperative positive SLN total tumor load (TTL) obtained from the OSNA assay and to determine whether this TTL predicts non-SLN metastasis in patients with clinically node-negative early-stage breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed invasive breast carcinoma
* Stage T1-3,N0 evaluated by physical exam or imaging according to AJCC v.7 and best clinical local practices
* Intraoperative evaluation of sentinel lymph node (SLN) by OSNA
* Complete dissection of axillary lymph nodes after the evaluation of the SLNs by OSNA
* Pathology report of the tumor and dissected lymph nodes that includes the following information:

  * primary tumor size (mm), tumor grade (Scarff-Bloom Richardson), estrogen receptor status
  * progesterone receptor status
  * HER2 status (ASCO/CAP guidelines)
  * Ki67 index
  * presence/absence of lymphovascular invasion
  * total number of sentinel and non-sentinel lymph nodes dissected during surgery
  * total number of positive and negative sentinel and non-sentinel lymph nodes, *size of the metastasis in both sentinel and non-sentinel lymph nodes
  * total tumoral load in each sentinel lymph node, expressed as number of CK19 mRNA copies per microliter.

Exclusion Criteria:

* Patients who underwent neoadjuvant chemotherapy
* CK19-negative breast tumor
* ALND with <10 lymph nodes
* In situ carcinoma only
* Metastatic breast cancer at time of diagnosis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cT1-3, N0 breast cancer, who had intraoperative SLN evaluation by OSNA assay with a complete axillary lymph node dissection.
Sampling Method: Non-Probability Sample
Enrollment: 701 (Actual)
Dates: Start 2012-06; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Estimate the negative predictive value of the technique OSNA. | At time of surgery
  Estimate the negative predictive value of the technique OSNA for the cutoff point that maximizes (tentatively, 10,000 to 15,000 copies / uL) of axillary lymph node involvement in breast cancer early N0.

SECONDARY OUTCOMES:
ROC curve that describes the assay | At time of surgery
  ROC curve (Receiver Operating Characteristic) from the true and false positives and negatives of OSNA test for different cutoffs
Sensitivity of the assay | At time of surgery
  Probability that OSNA in sentinel lymph nodes (SLN) is positive given that there is involvement of non-sentinel lymph nodes (NSLN)
Specificity of the assay | At time of surgery
  Probability that OSNA in SLN is negative because there is no involvement of NSLN
Likelihood ratio for the cutoff of 10,000-15,000 copies/uL | At time of surgery
  Likelihood ratio of positive and negative results
Positive predictive value at the cutoff of 10.000-15.000 copies/μL. | At time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Peg, MD, Principal Investigator — Vall d´Hebron University Hospital; Isabel Rubio, MD, PhD, Study Chair — Vall d´Hebron University Hospital; Martin Espinosa-Bravo, MD, PhD, Study Chair — Vall d´Hebron University Hospital
Locations (9):
- Spain (9):
  - Hospital Clínico Universitario de Santiago de Compostela, A Coruña
  - Hospital Universitario de Bellvitge, Barcelona
  - Vall d´Hebron University Hospital, Barcelona
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville
  - Instituto Valenciano de Oncología, Valencia

REFERENCES:
- [Result] Peg V, Espinosa-Bravo M, Vieites B, Vilardell F, Antunez JR, de Salas MS, Delgado-Sanchez JJ, Pinto W, Gozalbo F, Petit A, Sansano I, Del Mar Tellez M, Rubio IT. Intraoperative molecular analysis of total tumor load in sentinel lymph node: a new predictor of axillary status in early breast cancer patients. Breast Cancer Res Treat. 2013 May;139(1):87-93. doi: 10.1007/s10549-013-2524-z. Epub 2013 Apr 11. PMID 23576079
- [Result] Peg V, Espinosa-Bravo M, Vieites B, Vilardell F, Antúnez JJ, Salas MS, Sansano I, Delgado Sánchez JJ, Pinto W, Gozalbo F, Petit A, Rubio I. Intraoperative molecular analysis of sentinel lymph node as a new predictor of axillary status in early breast cancer. Poster session presented at: 35th Annual San Antonio Breast Cancer Symposium (SABCS); 2012 December 4th-8th; San Antonio, Texas, United States.
- See also: SOLTI Breast Cancer Research Group — http://www.gruposolti.org